CLINICAL TRIAL: NCT01358526
Title: A Randomized, Double-blind, Placebo-controlled, Multicenter Trial With an Enriched Study Design to Assess the Efficacy and Safety of Oxycodone/Naloxone Controlled-release Tablets (OXN) Compared to Placebo in Opioid-experienced Subjects With Moderate to Severe Pain Due to Chronic Low Back Pain Who Require Around-the-clock Opioid Therapy
Brief Title: Efficacy and Safety of Oxycodone/Naloxone Controlled-release Tablets (OXN) Compared to Placebo in Opioid-experienced Subjects With Moderate to Severe Chronic Low Back Pain
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Purdue Pharma LP (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ONU3701
Record Dates: First submitted 2011-05-20; First posted 2011-05-23 (Estimated); Results first posted 2014-09-03 (Estimated); Last update posted 2015-11-11 (Estimated); Status verified 2015-10

CONDITIONS: Low Back Pain
Keywords: Low back pain; Chronic pain; Opioid; Moderate to severe chronic low back pain
MeSH Terms: conditions — Low Back Pain; Chronic Pain | interventions — Oxycodone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- OXN (Experimental): Oxycodone/Naloxone Controlled-release Tablets (OXN)
  Interventions: Drug: Oxycodone/Naloxone Controlled-release
- Placebo (Placebo Comparator): Placebo tablets to match OXN
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Oxycodone/Naloxone Controlled-release — Oxycodone/Naloxone Controlled-release tablets (10/5 mg, 20/10 mg, 30/15 mg, 40/20 mg) taken orally every 12 hours
  Other Names: TARGINIQ ER
  Arms: OXN
Drug: Placebo — Placebo tablets to match OXN taken orally every 12 hours
  Arms: Placebo

SUMMARY:
The primary objective of this study is to assess the efficacy and safety of OXN compared to placebo in opioid-experienced subjects with moderate to severe pain due to chronic low back pain who require around-the-clock opioid therapy.

ELIGIBILITY:
Inclusion Criteria include:

* Male and female subjects ≥ 18 years of age with moderate to severe, chronic low back pain (lasting at least several hours daily) as their predominant pain condition for at least 3 months prior to screening period;
* The back pain must be related to nonmalignant and nonneuropathic conditions and without radiation or with only proximal radiation (above the knee);
* Subjects must be on opioid analgesic therapy for low back pain which:
* Has been ongoing for at least 4 weeks prior to the screening visit and,
* Consists of a stable opioid regimen at a total average daily dose equivalent to 20 to 160 mg (inclusive) of morphine for the last 2 weeks prior to the screening visit. Subjects taking tramadol ≥ 100 mg daily on a stable regimen for the last 2 weeks prior to the screening visit will also meet this criterion;
* Subjects must require continuation of opioid analgesic treatment in the range of 40 to 160 mg (inclusive) of morphine or its equivalent daily and be likely to benefit from chronic around-the-clock opioid therapy for the duration of the study;
* Subjects must have an average pain over the last 14 days score ≥ 5 (on an 11-point numerical rating scale [NRS]) at the screening visit, on their current opioid analgesic medication and, if applicable, nonopioid medication;
* Subjects must have an average pain over the last 24 hours score ≥ 5 (on an 11-point NRS) at the screening visit, on their current opioid analgesic medication and, if applicable, nonopioid medication;
* Subjects must be willing and able to be compliant with the protocol, capable of subjective evaluation, able to read and understand questionnaires, willing and able to use a diary per protocol, and read, understand, and sign the written informed consent in English.

Exclusion Criteria include:

* Female subjects who are pregnant (positive serum beta human chorionic gonadotropin [β hCG] test) or lactating;
* Subjects with any contraindication or any history of hypersensitivity to oxycodone, naloxone, or other opioids. This does not include subjects who have experienced common opioid side effects (e.g., nausea, constipation);
* Subjects with acute spinal cord compression, acute compression fracture, seronegative spondyloarthropathy, acute nerve root compression, cauda equina compression, fibromyalgia, reflex sympathetic dystrophy or causalgia (complex regional pain syndrome), diabetic amyotrophy, meningitis, discitis, or back pain due to secondary infection, tumor, or postherpetic neuralgia;
* Subjects with gout, unless controlled on stable suppressive treatment with colchicine or uric-acid-lowering therapy without any attacks for ≥ 2 years and the subject has not been using nonsteroidal anti-inflammatory drugs (NSAIDs) or COX-2 inhibitors on a regular basis;
* Subjects with pseudogout, psoriatic arthritis, active Lyme disease, rheumatoid arthritis or other inflammatory arthritis, or neuropathic pain conditions;
* Subjects who had surgical procedures directed towards the source of chronic low back pain within 6 months of the screening visit or planned during the study;
* Subjects with a history of opioid, alcohol, medication, or illicit drug abuse or addiction;
* Subjects who have received any investigational medication within 30 days of first dose of study drug;
* Subjects currently taking, or who have taken naloxone, naltrexone, methylnaltrexone, or alvimopan within 10 days before the screening visit;
* Subjects who have received study drug in a clinical study of oxycodone/naloxone controlled-release (OXN or ONU).

Other protocol specific inclusion/exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1095 (Actual)
Dates: Start 2011-05; Primary Completion 2012-10 (Actual); Study Completion 2012-11 (Actual)

CONTACTS AND LOCATIONS:
Locations (151):
- United States (151):
  - Alabama Orthopaedic Center, PC, Birmingham, Alabama
  - Alliance Clinical Research, Birmingham, Alabama
  - Winston Technology Research, LLC, Haleyville, Alabama
  - Monte Sano Clinical Research, LLC, Huntsville, Alabama
  - Research Facility, Mobile, Alabama
  - Radiant Research, Inc., Chandler, Arizona
  - Dedicated Clinical Research, Phoenix, Arizona
  - Arizona Research Center, Phoenix, Arizona
  - Clinical Research Advantage, Inc./Tatum Highlands Medical Associates, PLLC, Phoenix, Arizona
  - Quality of Life Medical & Research Center, LLC, Tucson, Arizona
  - Ortho Surgeons, Little Rock, Arkansas
  - Orange County Research Institute, Anaheim, California
  - Physician Alliance Research Center, Anaheim, California
  - Advanced Pain Research Institute, Arcadia, California
  - Southbay Pharma Research, Buena Park, California
  - Providence Clinical Research, Burbank, California
  - Med Center, Carmichael, California
  - Advanced Pain Management and Rehabilitation Medical Group, Inc., Castro Valley, California
  - Catalina Research Institute, LLC, Chino, California
  - Synergy Clinical Research of Escondido, Escondido, California
  - Valley Research, Fresno, California
  - RX Clinical Research, Inc., Garden Grove, California
  - TriWest Research Associates, La Mesa, California
  - Pacific Coast Pain Management Center, Laguna Hills, California
  - South Orange County Surgical Medical Group, Laguna Hills, California
  - Clinical Trials Research, Lincoln, California
  - L.A. Pain and Wellness Institute, Los Angeles, California
  - Newport Beach Clinical Research Associates, Inc., Newport Beach, California
  - Lotus Clinical Research, Pasadena, California
  - Northern California Clinical Research Center, Redding, California
  - Probe Clinical Research Corporation, Riverside, California
  - Northern California Research, Sacramento, California
  - Probe Clinical Research Corporation, Santa Ana, California
  - Denver Internal Medicine Group, Denver, Colorado
  - Front Range Clinical Research, Wheat Ridge, Colorado
  - New England Research Associates, LLC, Trumbull, Connecticut
  - Orthopedic Research Institute, Boynton Beach, Florida
  - Coastal Orthopedics & Pain Management, Bradenton, Florida
  - Southeast Clinical Research, LLC, Chiefland, Florida
  - Innovative Research of West Florida, Inc., Clearwater, Florida
  - Clinical Research of West Florida, Inc., Clearwater, Florida
  - Omega Research Consultants, LLC, DeBary, Florida
  - S & W Clinical Research, Fort Lauderdale, Florida
  - Southeastern Integrated Medical, PL, Gainesville, Florida
  - Health Care Family Rehab & Research Center, Hialeah, Florida
  - Eastern Research, Inc., Hialeah, Florida
  - Southeast Clinical Research, LLC, Jacksonville, Florida
  - Florida Institute of Medical Research, Jacksonville, Florida
  - Drug Study Institute, Jupiter, Florida
  - Pharma Care Research, Inc., Miami, Florida
  - Advanced Pharma CR, LLC, Miami, Florida
  - Compass Research, LLC, Orlando, Florida
  - Peninsula Research, Inc., Ormond Beach, Florida
  - Sarasota Clinical Research, LLC, Sarasota, Florida
  - Sarasota Pain Medicine Research, Sarasota, Florida
  - Vita Research Solutions & Medical Center, Inc., Tamarac, Florida
  - Stedman Clinical Trials, Tampa, Florida
  - Advanced Research Institute, Inc., Trinity, Florida
  - Palm Beach Research Center, West Palm Beach, Florida
  - National Pain Research Institute, LLC, Winter Park, Florida
  - Independent Neurodiagnostic Clinic, Atlanta, Georgia
  - In-Quest Medical Research, LLC, Duluth, Georgia
  - Georgia Institute for Clinical Research, LLC, Marietta, Georgia
  - Research Facility, Marietta, Georgia
  - Better Health Clinical Research, Inc., Newnan, Georgia
  - SouthCoast Medical Group, Savannah, Georgia
  - Georgia Clinical Research, LLC, Snellville, Georgia
  - The Pain Center, Boise, Idaho
  - Clinical Investigation Specialists, Inc., Gurnee, Illinois
  - Destiny Clinical Research, LLC, Evansville, Indiana
  - MediSphere Medical Research Center, LLC, Evansville, Indiana
  - Northwest Indiana Center for Clinical Research, Valparaiso, Indiana
  - International Clinical Research Institute, Inc., Leawood, Kansas
  - Clinical Trials Technology, Inc. CTT Consultants, Inc., Prairie Village, Kansas
  - The Pain Treatment Center of the Bluegrass, Lexington, Kentucky
  - Louisiana Research Associates, Inc., New Orleans, Louisiana
  - Research Facility, New Orleans, Louisiana
  - Mid-Atlantic Medical Research Centers, Hollywood, Maryland
  - MidAtlantic Pain Medicine Center, Pikesville, Maryland
  - Beacon Clinical Research, LLC, Brockton, Massachusetts
  - ActivMed Practices and Research, Haverhill, Massachusetts
  - Medvadis Research Corporation, Watertown, Massachusetts
  - Great Lakes Research Group, Inc., Bay City, Michigan
  - Great Lakes Family Care, Cadillac, Michigan
  - Great Lakes Research Group, Inc., Pinconning, Michigan
  - Medex Healthcare Research, Inc., St Louis, Missouri
  - Mercy Health Research, St Louis, Missouri
  - Sundance Clinical Research, LLC, St Louis, Missouri
  - Meridian Clinical Research, LLC, Omaha, Nebraska
  - Research Facility, Las Vegas, Nevada
  - South Jersey Medical Associates, P.A., Blackwood, New Jersey
  - University of Medicine & Dentistry of New Jersey - School of Osteopathic Medicine (UMDNJ), Stratford, New Jersey
  - Five Towns Neuroscience Research/Five Towns Neurology, Cedarhurst, New York
  - Long Island Gastrointestinal Research Group, LLP, Great Neck, New York
  - Medex Healthcare Research, Inc., New York, New York
  - Research Across America, New York, New York
  - Upstate Clinical Research Associates, LLC, Williamsville, New York
  - Gaffney Health Services, Charlotte, North Carolina
  - Box Arthritis & Rheumatology of the Carolinas, PLLC, Charlotte, North Carolina
  - PharmQuest, Greensboro, North Carolina
  - Peters Medical Research, High Point, North Carolina
  - Plains Medical Clinic, LLC, Fargo, North Dakota
  - Clinical Inquest Center Ltd., Beavercreek, Ohio
  - Community Research, Cincinnati, Ohio
  - Columbus Clinical Research, Inc., Columbus, Ohio
  - Hometown Urgent Care and Research, Dayton, Ohio
  - Prestige Clinical Research, Franklin, Ohio
  - Hometown Urgent Care and Research, Springfield, Ohio
  - J L Clinical Research, Tiffin, Ohio
  - Bone Joint and Spine Surgeons, Inc., Toledo, Ohio
  - Pharmacotherapy Research Associates, Inc., Zanesville, Ohio
  - Neuropsychiatric Center and NPC Research, Oklahoma City, Oklahoma
  - Health Research Institute, Oklahoma City, Oklahoma
  - Paradigm Research Professionals, LLC, Oklahoma City, Oklahoma
  - Bend Memorial Clinic, Bend, Oregon
  - Pain Consultants of Oregon, Eugene, Oregon
  - Willamette Valley Clinical Studies, Eugene, Oregon
  - Sunstone Medical Research, LLC, Medford, Oregon
  - Allegheny Pain Management, PC, Altoona, Pennsylvania
  - Paramount Clinical Research, Bridgeville, Pennsylvania
  - Altoona Center for Clinical Research, Duncansville, Pennsylvania
  - The Clinical Trial Center, LLC, Jenkintown, Pennsylvania
  - Central Pennsylvania Clinical Research, Mechanicsburg, Pennsylvania
  - CRI Worldwide, LLC, Philadelphia, Pennsylvania
  - Dairyland Medical Center, Red Lion, Pennsylvania
  - New England Center for Clinical Research, Inc, Cranston, Rhode Island
  - Hartwell Research Group, LLC, Anderson, South Carolina
  - Greenville Pharmaceutical Research, Inc., Greenville, South Carolina
  - Internal Medicine of Greer, Greer, South Carolina
  - Meridian Clinical Research, Dakota Dunes, South Dakota
  - Health Concepts Wellness Center, Rapid City, South Dakota
  - Integrity Clinical Research, LLC, Huntingdon, Tennessee
  - FutureSearch Trials of Neurology, Austin, Texas
  - Austin Center for Clinical Research, Austin, Texas
  - Corpus Christi Pain Medicine, Corpus Christi, Texas
  - FutureSearch Trials of Dallas, Dallas, Texas
  - Pineloch Medical Clinic, Houston, Texas
  - Clinical Trial Network, Houston, Texas
  - Southwest Clinical Trials, Houston, Texas
  - Protenium Clinical Research, LLC, Hurst, Texas
  - TEAM Research of Central Texas, Killeen, Texas
  - West Texas Medical Associates, San Angelo, Texas
  - Sun Research Institute, San Antonio, Texas
  - Research Facility, Bountiful, Utah
  - Summit Pain Management, Murray, Utah
  - Alpine Medical Group, Salt Lake City, Utah
  - Highland Clinical Research, Salt Lake City, Utah
  - Virginia Research Center, Midlothian, Virginia
  - Hilltop Medical Center, Virginia Beach, Virginia
  - Independence Family Medicine, Virginia Beach, Virginia
  - Universal Research Group, Tacoma, Washington

REFERENCES:
- See also: TARGINIQ ER Labeling — http://www.accessdata.fda.gov/drugsatfda_docs/label/2014/205777lbl.pdf

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First subject first visit: 25-May-2011; Last subject last visit: 15-Oct-2012. The study was conducted at 132 medical/research sites in the United States.
Pre-assignment Details: Opioid-experienced subjects with moderate to severe pain due to chronic low back pain, who required around-the-clock opioid therapy.
Groups:
- Open-label Titration OXN: The open-label titration was designed to identify a stable, effective, and tolerable dose of OXN for each subject.
- OXN Group: Oxycodone/Naloxone Controlled-release Tablets (OXN)
  Oxycodone/Naloxone Controlled-release: Oxycodone/Naloxone Controlled-release tablets (10/5 mg, 20/10 mg, 30/15 mg, 40/20 mg) taken orally every 12 hours
- Placebo Group: Placebo tablets to match OXN
  Placebo: Placebo tablets to match OXN taken orally every 12 hours
Period: Open-label Titration Period
Arm/Group | Open-label Titration OXN | OXN Group | Placebo Group
Started | 1095 | 0 | 0
Completed | 601 (1 subject was randomized but never received double-blind treatment: Randomized Safety Population=600) | 0 | 0
Not Completed | 494 | 0 | 0
Not completed — Adverse Event | 95 | 0 | 0
Not completed — Withdrawal by Subject | 65 | 0 | 0
Not completed — Lost to Follow-up | 25 | 0 | 0
Not completed — Lack of Efficacy | 107 | 0 | 0
Not completed — Confirmed or suspected diversion | 16 | 0 | 0
Not completed — Administrative | 8 | 0 | 0
Not completed — Did not qualify | 178 | 0 | 0
Period: Double-blind Phase
Arm/Group | Open-label Titration OXN | OXN Group | Placebo Group
Started | 0 | 298 (1 subject was randomized but never received double-blind treatment: Randomized Safety Population=600) | 302 (1 subject was randomized but never received double-blind treatment: Randomized Safety Population=600)
Completed | 0 | 218 | 181
Not Completed | 0 | 80 | 121
Not completed — Adverse Event | 0 | 24 | 23
Not completed — Withdrawal by Subject | 0 | 10 | 8
Not completed — Lost to Follow-up | 0 | 4 | 1
Not completed — Lack of Efficacy | 0 | 31 | 73
Not completed — Confirmed or suspected diversion | 0 | 5 | 6
Not completed — Administrative | 0 | 6 | 10

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | OXN Group | Placebo Group | Total
Number analyzed (Participants) | 298 | 302 | 600
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.5 (11.69) | 53.0 (10.97) | 53.2 (11.33)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 162 | 176 | 338
  Male | 136 | 126 | 262
Race/Ethnicity, Customized [Number; unit: participants]
  White | 229 | 233 | 462
  Black or African American | 53 | 61 | 114
  Asian | 8 | 3 | 11
  American Indian or Alaska Native | 1 | 3 | 4
  Other | 7 | 2 | 9

OUTCOME MEASURES:

1. Primary Outcome: The "Average Pain Over the Last 24 Hours" at Week 12 of the Double-blind Period
Description: The "average pain over the last 24 hours" score was collected using an 11-point numerical rating scale ranging from 0 to 10; where 0=no pain and 10=pain as bad as you can imagine.
Time Frame: 24 hours (Week 12)
Population: The full analysis population for efficacy (N = 600) was the group of subjects who were randomized and received at least 1 dose of double-blind study drug
Measure: Mean (Standard Error); unit: units on a scale (0 - 10)
Arm/Group | OXN Group | Placebo Group
Number analyzed (Participants) | 298 | 302
units on a scale (0 - 10) | 3.86 (0.116) | 4.32 (0.115)
Statistical Analysis 1: Comparison: OXN Group vs Placebo Group; Test type: Superiority or Other; p = 0.0055, Mixed Models Analysis — A gate-keeping strategy and a Bonferroni-Holm method was used to control the family-wise (primary and secondary efficacy analysis) error rate at the 5% level; Mixed-model repeated measures analysis of pain data using a pattern mixture model framework; Mean Difference (Final Values) = 0.45, 95% CI 2-sided [0.13 to 0.77], Standard Error of Mean 0.163

2. Secondary Outcome: The Sleep Disturbance Subscale of the MOS Sleep Scale at Weeks 4, 8, and 12
Description: The scale consists of 12 individual items (4 sleep disturbance, 2 sleep adequacy, 1 quantity of sleep, 3 somnolence, 1 snoring, 1 shortness of breath). Only Sleep Disturbance Subscale questions 1, 3, 7, and 8 were analyzed; scores range from 0 to 100, where higher scores indicate greater sleep disturbance.
Time Frame: Weeks 4, 8, and 12
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | OXN Group | Placebo Group
Number analyzed (Participants) | 298 | 302
units on a scale
  Week 4 | 32.5 [29.4 to 35.7] | 38.0 [34.8 to 41.3]
  Week 8 | 30.8 [27.8 to 33.9] | 36.8 [33.6 to 39.9]
  Week 12 | 31.1 [28.1 to 34.2] | 36.4 [33.2 to 39.7]
Statistical Analysis 1: Comparison: OXN Group vs Placebo Group; Test type: Superiority or Other; p = 0.0191, Mixed Models Analysis; Mixed-model repeated measures analysis; Mean Difference (Final Values) = 5.3, 95% CI 2-sided [0.9 to 9.8], Standard Error of Mean 2.26 — Mean difference (final values) is the treatment comparison estimated using mixed model repeated measures analysis with effect for treatment, time (weeks 4, 8, 12), treatment by time interaction, and prerandomization value. Subject is a random effect

3. Secondary Outcome: Patient Global Impression of Change (PGIC)
Description: The PGIC observational scale was completed by the subject. Subjects were asked to assess the change in overall status relative to the start of the study. The scale has only 1 item, which measures global change of overall status by the subject on a 7-point scale (Very much improved, Much improved, Minimally improved, No change, Minimally worse, Much worse, Very much worse), where 1 = very much improved and 7 = very much worse. The proportion of subjects responding "much improved" and "very much improved" was summarized by treatment group and compared between groups using an exact test.
Time Frame: Week 12
Population: as for outcome 1
Measure: Number; unit: participants (responders)
Arm/Group | OXN Group | Placebo Group
Number analyzed (Participants) | 298 | 302
participants (responders) | 153 | 109
Statistical Analysis 1: Comparison: OXN Group vs Placebo Group; Test type: Superiority or Other; p = 0.0002, Fisher Exact — The proportion of subjects responding "much improved" and "very much improved" was summarized by treatment group and compared between groups using an exact test

4. Other Pre Specified Outcome: Responder Analysis for Subjects With a ≥ 30% Reduction in Pain Compared to Baseline
Description: A subject's response to treatment was defined as the percentage reduction from the screening mean pain score to the "average pain over the last 24 hours" score for week 12 of the double-blind period.
Time Frame: Week 12
Population: as for outcome 1
Measure: Number; unit: participants (responders)
Arm/Group | OXN Group | Placebo Group
Number analyzed (Participants) | 298 | 302
participants (responders) | 164 | 124
Statistical Analysis 1: Comparison: OXN Group vs Placebo Group; Proportion of subjects with a response to treatment that is ≥ 30%; Test type: Superiority or Other; p = 0.0006, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel test: responder as dependent variable, treatment as explanatory variable, dose at time of randomization as stratifying factor

5. Other Pre Specified Outcome: Responder Analysis for Subjects With a ≥ 50% Reduction in Pain Compared to Baseline
Description: as for outcome 4
Time Frame: Week 12
Population: as for outcome 1
Measure: Number; unit: participants (responders)
Arm/Group | OXN Group | Placebo Group
Number analyzed (Participants) | 298 | 302
participants (responders) | 109 | 75
Statistical Analysis 1: Comparison: OXN Group vs Placebo Group; Proportion of subjects with a response to treatment that is ≥ 50%; Test type: Superiority or Other; p = 0.0018, Cochran-Mantel-Haenszel; [statistical method as in outcome 4, analysis 1]

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were reported from start of study participation through the period beyond study completion.
Description: AEs were learned of through spontaneous reports and/or subject interview, or were observed during physical examinations or other safety assessments. Ongoing AEs were followed until resolution or 30 days after last study drug dose. Serious AEs up to 30 days following the last study visit were followed until the AE or sequelae resolved or stabilized.
Groups:
- Open-label Titration OXN; Double-blind OXN: Oxycodone/Naloxone Controlled-release Tablets (OXN)
  Oxycodone/Naloxone Controlled-release: Oxycodone/Naloxone Controlled-release tablets (10/5 mg, 20/10 mg, 30/15 mg, 40/20 mg) taken orally every 12 hours
- Double-blind Placebo: Placebo tablets to match OXN
  Placebo: Placebo tablets to match OXN taken orally every 12 hours
Arm/Group | Open-label Titration OXN | Double-blind Placebo | Double-blind OXN
Serious Adverse Events (participants affected / at risk) | 11/1095 | 12/302 | 19/298
Other Adverse Events (participants affected / at risk) | 79/1095 | 34/302 | 41/298
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Open-label Titration OXN (N=1095) | Double-blind Placebo (N=302) | Double-blind OXN (N=298)
Acute myocardial infarction (Cardiac disorders) | 0 | 2 | 0
Angina pectoris (Cardiac disorders) | 0 | 0 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 1
Non-cardiac chest pain (General disorders) | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 1
Impaired gastric emptying (Gastrointestinal disorders) | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 0 | 0
Oesophageal stenosis (Gastrointestinal disorders) | 1 | 0 | 0
Rectal perforation (Gastrointestinal disorders) | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 0 | 1
Cholecystitis acute (Hepatobiliary disorders) | 0 | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 1 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 1
Gallbladder empyema (Infections and infestations) | 0 | 1 | 0
Gangrene (Infections and infestations) | 0 | 1 | 0
Ludwig angina (Infections and infestations) | 0 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 1 | 1
Gun shot wound (Injury, poisoning and procedural complications) | 0 | 1 | 0 — Death
Overdose (Injury, poisoning and procedural complications) | 1 | 0 | 0
Drug screen positive (Investigations) | 5 | 1 | 9
Hepatic enzyme increased (Investigations) | 0 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Systemic lupus erythematosus (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Syncope (Nervous system disorders) | 0 | 0 | 1
Drug abuse (Psychiatric disorders) | 3 | 0 | 0
Renal failure (Renal and urinary disorders) | 0 | 1 | 0
Substance abuse (Social circumstances) | 0 | 2 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Open-label Titration OXN (N=1095) | Double-blind Placebo (N=302) | Double-blind OXN (N=298)
Nausea (Gastrointestinal disorders) | 79 | 14 | 25
Drug screen positive (Investigations) | 23 | 20 | 19

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days